CLINICAL TRIAL: NCT02963116
Title: A Randomized, 5-Period, 5-Treatment, Single-Dose, Open-Label, Single-Center, Crossover Study to Estimate the Effect of AZD5718 on the Pharmacokinetics of Rosuvastatin, and to Assess the Relative Bioavailability of AZD5718 Oral Suspension vs AZD5718 IR Tablet Formulation and the Food Effect of AZD5718.
Brief Title: A Study to Estimate the Effect of AZD5718 on the Pharmacokinetics (What Does the Body Does to the Drug) of Rosuvastatin to Measure the Relative Bioavailability (the Extent to Which a Drug or Other Substance Becomes Available to the Body) of AZD5718 Oral Suspension vs AZD5718 Immediate Release Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: D7550C00002
Record Dates: First submitted 2016-11-04; First posted 2016-11-15 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: High Risk Coronary Artery Disease
Keywords: Pharmacokinetics (PK); Bioavailability (BA); Safety; Tolerability; Healthy Volunteers
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment A (Experimental): 10 mg rosuvastatin tablet alone (fasting state)
  Interventions: Drug: Rosuvastatin tablet
- Treatment B (Experimental): 10 mg rosuvastatin tablet + 200 mg of AZD5718 IR tablet (2 x 100 mg tablet) (fasting state)
  Interventions: Drug: AZD5718 IR tablet; Drug: Rosuvastatin tablet
- Treatment C (Experimental): 200 mg of AZD5718 IR tablet (2 x 100 mg tablet) (fasting state)
  Interventions: Drug: AZD5718 IR tablet
- Treatment D (Experimental): 200 mg of AZD5718 oral suspension 50 mg/mL (fasting state)
  Interventions: Drug: AZD5718 oral suspension
- Treatment E (Experimental): 200 mg of AZD5718 IR tablet (2 x 100 mg tablet) (fed state)
  Interventions: Drug: AZD5718 IR tablet

INTERVENTIONS:
Drug: AZD5718 IR tablet
  Arms: Treatment B; Treatment C; Treatment E
Drug: AZD5718 oral suspension
  Arms: Treatment D
Drug: Rosuvastatin tablet
  Arms: Treatment A; Treatment B

SUMMARY:
This study is a randomized, open-label, 5-period, 5-treatment, single-dose, single-center, crossover study to estimate the effect of AZD5718 on the pharmacokinetics (PK) of rosuvastatin, and to assess the relative bioavailability of AZD5718 oral suspension vs AZD5718 immediate release (IR) Tablet Formulation and the Food Effect of AZD5718 in Healthy Volunteers. The study will be performed at a single study center.

DETAILED DESCRIPTION:
The study will comprise:

* A Screening period of maximum 28 days;
* Five treatment periods during which subjects will be resident from the morning on the day before dosing with the IMP (Day -1) until at least 48 hours after dosing; discharge will be on the morning of Day 3, and
* A Follow-up Visit within 7 to 10 days after the last administration of the IMPs.
* There will be a minimum of a 7 days washout between each treatment period.

Each subject will receive 5 treatments. The following treatments will be given:

* Treatment A: 10 mg rosuvastatin tablet alone (fasting state)
* Treatment B: 10 mg rosuvastatin tablet + 200 mg of AZD5718 IR tablet (2 x 100 mg tablet) (fasting state)
* Treatment C: 200 mg of AZD5718 IR tablet (2 x 100 mg tablet) (fasting state)
* Treatment D: 200 mg of AZD5718 oral suspension 50 mg/mL (fasting state)
* Treatment E: 200 mg of AZD5718 IR tablet (2 x 100 mg tablet) (fed state)

Each subject will be involved in the study for approximately 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, subjects should fulfill the following criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male and/or female subjects (of non childbearing potential) aged 18 to 50 years (inclusive) with suitable veins for cannulation or repeated venipuncture.
3. Females must have a negative pregnancy test at the Screening Visit and on admission to the unit, must not be lactating and must be of non-childbearing potential, confirmed at the Screening Visit by fulfilling one of the following criteria 3.1. Postmenopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle stimulating hormone levels in the postmenopausal range.

   3.2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral ophorectomy or bilateral salpingectomy but excluding bilateral tubal ligation.
4. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg, inclusive.
5. Provision of signed, written and dated informed consent for optional genetic/biomarker research. If a subject declines to participate in the genetic component of the study, there will be no penalty or loss of benefit to the subject. The subject will not be excluded from other aspects of the study.

Exclusion Criteria:

Subjects will not enter the study if any of the following exclusion criteria are fulfilled:

1. History of any clinically significant disease or disorder which, in the opinion of the PI, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
4. Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, at the Screening Visit and/or admission to the study unit as judged by the PI including: - Aminotransferase (ALT) > upper limit of normal (ULN); - Aspartate aminotransferase (AST) > ULN; - Total bilirubin (TBL) > ULN; and - Gamma glutamyl transpeptidase (GGT) > ULN.
5. Any clinically significant abnormal findings in vital signs at the Screening Visit and/or admission to the study unit, as judged by the PI defined as any of the following: - Systolic BP (SBP) < 90 mmHg or ≥ 140 mmHg; - Diastolic BP (DBP) < 50 mmHg or ≥ 90 mmHg; and - Pulse < 45 or > 85 beats per minute (bpm).
6. Any clinically significant abnormalities (at the Screening Visit and admission) in rhythm, conduction or morphology of the resting ECG and any clinically significant abnormalities in the 12-lead ECG, as considered by the investigator that may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology, particularly in the protocol defined primary lead or left ventricular hypertrophy.
7. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
8. Subjects with myopathy.
9. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or 1 month after the last visit whichever is the longest. Note: subjects consented and screened, but not randomized in this study or a previous phase I study, are not excluded.
10. Plasma donation within 1 month of the Screening Visit or any blood donation/loss more than 500 mL during the 3 months prior to the Screening Visit.
11. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to AZD5718 and/or rosuvastatin.
12. Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 3 months prior to the Screening Visit.
13. Positive screen for drugs of abuse or cotinine at the Screening Visit or on each admission to the study center or positive screen for alcohol on each admission to the study center.
14. Excessive intake of caffeine containing drinks or food (e.g., coffee, tea, chocolate), as judged by the investigator.
15. Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
16. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life. Note: Hormonal replacement therapy is not allowed for females.
17. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the PI.
18. Involvement of any AstraZeneca, PAREXEL or study site employee or their close relatives. 19. Subjects who have previously received AZD5718.

20. Judgment by the PI that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.

21. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order In addition, the following is considered a criterion for the exclusion from the optional genetic component of the study: 22. Previous bone marrow transplant. 23. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection or previous bone marrow transplant.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from time zero to infinity (AUC) of Rosuvastatin | Pre-dose, and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 h post-dose
  Assessment of AUC of rosuvastatin when administered alone and in combination with AZD5718 in healthy volunteers.
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-last)] of Rosuvastatin | Pre-dose, and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 h post-dose
  Assessment of AUC(0-last) of rosuvastatin when administered alone and in combination with AZD5718 in healthy volunteers.
Maximum observed plasma concentration (Cmax) of Rosuvastatin | Pre-dose, and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 h post-dose
  Assessment of Cmax of rosuvastatin when administered alone and in combination with AZD5718 in healthy volunteers.

SECONDARY OUTCOMES:
Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t½) of Rosuvastatin - | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 h post-dose. (Only Treatment A and B)
  Assessment of t½ of rosuvastatin.
Time to reach maximum observed plasma concentration (tmax) of rosuvastatin | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 h post-dose. (Only Treatment A and B)
  Assessment of tmax of rosuvastatin.
AUC of AZD5718 | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 h post-dose (Only Treatment B, C, D, and E)
  Assessment of AUC of AZD5718.
AUC(0-last) of AZD5718 | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 h post-dose (Only Treatment B, C, D, and E)
  Assessment of AUC(0-last) of AZD5718.
Cmax of AZD5718 | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 h post-dose (Only Treatment B, C, D, and E)
  Assessment of Cmax of AZD5718.
tmax of AZD5718 | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 h post-dose (Only Treatment B, C, D, and E)
  Assessment of tmax of AZD5718.
t½ of AZD5718 | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 h post-dose (Only Treatment B, C, D, and E)
  Assessment of t½ of AZD5718.
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) of AZD5718 | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 h post-dose (Only Treatment B, C, D, and E)
  Assessment of CL/F of AZD5718.
Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) of AZD5718 | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 h post-dose (Only Treatment B, C, D, and E)
  Assessment of Vz/F of AZD5718.
Adverse events (AEs) | Screening, Day -1 and Days 1 to 3 (treatment periods 1 to 5) and follow up visit (7-10 days post final dose)
  Assessment of the safety in terms of the incidences of the AEs.
Vital signs (systolic and diastolic blood pressure, pulse rate and body temperature) | Screening, Day -1, Pre-dose, 48 h post-dose and Follow-up visit (7-10 days post final dose)
  Assessment of the safety in terms of the Vital signs (systolic and diastolic blood pressure, pulse rate).
Electrocardiogram (ECG) | Screening, Day -1, Pre-dose, 48 h post-dose and Follow-up visit (7-10 days post final dose)
  Assessment of the safety in terms of the ECG.
Physical examination | Screening, Day -1 (brief), 48 h (brief) post-dose
  Assessment of the safety in terms of the physical examination.
Laboratory assessments (hematology, clinical chemistry and urinalysis). | Screening, Day -1 (only limited clinical laboratory evaluations will be performed), Pre-dose, 48 h post-dose and Follow-up Visit (7-10 days post final dose)
  Assessment of the safety in terms of the Clinical laboratory assessments (hematology, clinical chemistry and urinalysis).

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Muna Albayaty, MBChB, MSc, MFPM, Principal Investigator — PAREXEL Early Phase Clinical Unit London
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- [Derived] Ericsson H, Nelander K, Heijer M, Kjaer M, Lindstedt EL, Albayaty M, Forte P, Lagerstrom-Fermer M, Skrtic S. Phase 1 Pharmacokinetic Study of AZD5718 in Healthy Volunteers: Effects of Coadministration With Rosuvastatin, Formulation and Food on Oral Bioavailability. Clin Pharmacol Drug Dev. 2020 Apr;9(3):411-421. doi: 10.1002/cpdd.756. Epub 2019 Dec 2. PMID 31793171